CLINICAL TRIAL: NCT06489886
Title: Nutrient and Hormonal Profile and Muscle Protein Synthesis Response to Consuming Chicken Grown Using Different Farming Practices
Brief Title: Nutrient and Hormonal Profile and Muscle Protein Synthesis Response to Consuming Chicken
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2190600
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Effect of Food
Keywords: Muscle protein Synthesis; post-prandial nutrient and hormonal profile; farming practices

STUDY DESIGN:
Intervention Model Description: Participants will consume a meal of chicken, which type (conventional vs. regenerative ) consumed will be randomized where neither the participant nor investigator will know which meal is being consumed. Each participant will repeat the protocol two times.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A randomized double-blind crossover design with neither the subjects nor the investigators knowing who is on which food. The interventions will be coded using a blinded alphabetical letter code (A, B). A delegate researcher (independent party not further involved in the study) will randomize all interventions using a computer-generated randomization list. The delegate will hand in the code-breaker to the principal investigator in a sealed envelope. The envelope will be stored in a locked filing cabinet in the principal investigator's office, which will also be locked when unoccupied. The envelope will be opened by the principal investigator after completing the analysis of blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Chicken (Experimental): This arm will be given a meal of 100 grams (~32g of protein) boneless-skinless conventional chicken breast meat together with 250mL of water
  Interventions: Other: Conventional Chicken
- Regenerative Chicken (Experimental): This arm will be given a meal of 100 grams (~32g of protein) boneless-skinless regenerative chicken breast meat together with 250mL of water
  Interventions: Other: Regenerative Chicken

INTERVENTIONS:
Other: Conventional Chicken — This arm will be given a meal of 100 grams (~32g of protein) boneless-skinless convential chicken breast meat together with 250mL of water
  Arms: Conventional Chicken
Other: Regenerative Chicken — This arm will be given a meal of 100 grams (~32g of protein) boneless-skinless regenerative chicken breast meat together with 250mL of water
  Arms: Regenerative Chicken

SUMMARY:
The study aims to evaluate if there is a difference between eating conventionally raised or organic chicken. The investigators will measure and compare the nutrient and hormone levels in the participant's blood and the muscle protein synthesis rate (the rate at which your body builds muscle) after eating chicken from different farming practices. This will help the investigators to understand if these farming practices impact muscle protein synthesis and overall health.

Specific aim 1: Describe the post-prandial nutrient and hormonal profile in serum in the 3 hours following consumption of 100 grams (~32g of protein) of boneless-skinless conventional vs. regenerative chicken breast meat.

Specific aim 2: Compare the ability of boneless-skinless chicken breasts grown with these two farming practices to activate mTORC1-specific and whole muscle protein synthesis in an in vitro model of muscle.

DETAILED DESCRIPTION:
Indicators of longevity in humans include skeletal muscle mass and strength. Muscle mass depends on the balance between myofibrillar protein synthesis and degradation, influenced by diet and physical activity. Muscle strength correlates with muscle mass, and weight lifting until failure increases muscle protein synthesis, enhancing muscle mass and strength over time. Protein intake is crucial for positive protein balance and muscle growth. Animal proteins promote muscle synthesis more effectively than plant proteins. Limited research exists on the impact of agricultural practices on meat quality. Studies indicate that organic meat may have higher nutritional value and better lipid profiles. This project aims to compare the serum nutrient, hormonal profiles, and muscle protein synthesis rates after consuming isonitrogenous amounts of chicken from conventional versus regenerative/organic practices.

The purpose of the study is to quantify and compare the serum nutrient and hormonal profile, and muscle protein synthesis rates, in response to consuming isonitrogenous amounts of chicken grown using different agricultural practices (conventional vs. regenerative)

Specific aim 1: Describe the post-prandial nutrient and hormonal profile in serum in the 3 hours following consumption of 100 grams (~32g of protein) of boneless-skinless conventional vs. regenerative chicken breast meat.

Specific aim 2: Compare the ability of boneless-skinless chicken breasts grown with these two farming practices to activate mTORC1-specific and whole muscle protein synthesis in an in vitro model of muscle.

Study participant will come to the CTSC Clinical Research Center on two separate occasions.

The two study visits will be scheduled over a 2-week period (i.e. once per week for 2 weeks), at the same time in the morning following an overnight (> 12-hour) fast. The participants will be asked to refrain from vigorous exercise, caffeine, nicotine and alcohol for 24 hours before each visit. Female participants will be asked to schedule their study visits within the first two weeks of their menstrual cycle (starting on the first day of menstrual bleeding), to control for ovarian hormone fluctuations which may impact digestion and metabolism.

Upon arrival at the research center on the first test visit, each participant's height and weight will be measured. Each participant will also fill out a questionnaire regarding physical activity and dietary habits.

I. Baseline blood draw.

Participants will then be placed in individual testing rooms, equipped with a reclining phlebotomy armchair. A registered nurse or nurse practitioner will insert a 22G catheter in a forearm vein and an initial 5 mL baseline blood sample will be collected.

II. Test meal.

After the baseline blood sample is collected, participants will consume one of the two chicken test meals. The meat will be equivalent to an isonitrogenous amount of 20 g of protein:

The food will be weighed before cooking and an eighth of a teaspoon of salt will be added for palatability. The boneless-skinless chicken breasts will be grilled on an indoor electric grill until the internal temperature reaches 165-170°F to comply with the USDA Recommendations for Food Safety (Chicken, minimum 165°F). The internal temperature of the chicken breasts will be determined using a meat thermometer. The chicken will be served to the participants as soon as it has finished cooking. Participants will be asked to consume each boneless-skinless chicken breast without condiments within a 10-minute period and instructed to chew thoroughly. Participants will also be asked to drink a 250 mL glass of water with the meal.

III. Postprandial blood draws.

Following consumption of the test meal, the participants will remain at the research site, in their individual testing room, for another 3 hours, they may bring books or electronic devices to pass the time. Five more blood samples of 5 mL each will be obtained at 30, 60, 90, 120 and 180 minutes after the test meal, totaling six blood draws of 5mL per visit (30mL per visit), and 60 mL of blood drawn in total for each subject completing the entire study.

Blood will be collected in 5 mL serum-separating tubes. The blood will be allowed to clot for before centrifugation at 1000 x g for 10 minutes. The serum will be frozen and kept at -80°C until processed. 1 milliliter of each serum sample will be used for determining nutrient and hormone concentrations. The rest of the serum will be used for muscle protein synthesis and mTORC1 bioassay analysis.

ELIGIBILITY:
Inclusion Criteria:

Healthy active males and females (To be considered active, volunteers must meet the following American College of Sports Medicine's guideline for physical activity for healthy adults: performing at least 150 minutes per week of moderate-to-vigorous intensity physical activity.

Age18-30 years

Normal weight (BMI between 18 and 25 kg/m2

Exclusion Criteria:

Health or dietary restrictions that would prevent consumption of the test foods

Known food allergy to chicken

Anemia (low red blood cell count)

Overweight or obesity (BMI > 25 kg/m2)

Receiving any medication that may interfere with the study

Metabolic or endocrine disorder that would affect the digestion, absorption, and/or physiological response to any of the nutrients ingested.

Currently not meeting the ACSM physical activity recommendations (IPAQ score < 150 min/week of moderate-to-vigorous physical activity.

Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
post-prandial amino acid profile | Baseline (0 hour) to 30, 60, 90, 120 and 180 minutes after consumed meal
  Serum samples are extracted with 1mL of modified Folch extraction, followed by vacuum centrifugation for drying. Dried samples will be reconstituted with 100 μl of 75% ACN/water. The supernatant is then injected into Aligent UPLC-QqQ for analysis of targeted free amino acids, short peptides, and other metabolites.
post-prandial short peptide profile | Baseline (0 hour) to 30, 60, 90, 120 and 180 minutes after consumed meal
  Serum samples are extracted with 1mL of modified Folch extraction, followed by vacuum centrifugation for drying. Dried samples will be reconstituted with 100 μl of 75% ACN/water. The supernatant is then injected into Aligent UPLC-QqQ for analysis of targeted free amino acids, short peptides, and other metabolites.
Muscle protein synthesis | Baseline (0 hour) to 30, 60, 90, 120 and 180 minutes after consumed meal
  To measure muscle protein synthesis, stably transfected C2C12 muscle cells with a plasmid (pcDNA3 luciferase) will be used. C2C12Luc cells will be plated in 24-well plates and differentiated over 4 days. Differentiated C2C12 cells will be fasted by washing with PBS and then treating them with Test Media (20% DMEM) for 15 minutes. Fasted muscle cells will then be treated with Test Media containing 10% baseline or fed serum (from blood samples at 30, 60, 90,120 and 180 minutes after meal) for 3 hours. Cells will be collected in passive lysis buffer and firefly luciferase activity will be determined.
mTORC1 specific protein synthesis | Baseline (0 hour) to 30, 60, 90, 120 and 180 minutes after consumed meal
  To measure the ability of meal of chicken (conventional or regenerative) to activate mTORC1, stably transfected C2C12 muscle cells with a plasmid (pcDNA3-TOP luciferase) where the luciferase mRNA contains a 5'TOP. 5'TOP mRNA, which specifically regulated by mTORC1 activity, will be used.
  Differentiated C2C12TOPLuc muscle cells in 24-well plates will be stimulated using the baseline or fed serum (from blood samples at 30, 60, 90,120 and 180 minutes after meal). The degree of mTORC1 activation will be determined as the difference in slopes between the baseline and fed sera.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Baar, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis CTSC Clinical Research Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruiz JR, Sui X, Lobelo F, Morrow JR Jr, Jackson AW, Sjostrom M, Blair SN. Association between muscular strength and mortality in men: prospective cohort study. BMJ. 2008 Jul 1;337(7661):a439. doi: 10.1136/bmj.a439. PMID 18595904
- [Background] Srikanthan P, Karlamangla AS. Muscle mass index as a predictor of longevity in older adults. Am J Med. 2014 Jun;127(6):547-53. doi: 10.1016/j.amjmed.2014.02.007. Epub 2014 Feb 18. PMID 24561114
- [Background] Schiaffino S, Dyar KA, Ciciliot S, Blaauw B, Sandri M. Mechanisms regulating skeletal muscle growth and atrophy. FEBS J. 2013 Sep;280(17):4294-314. doi: 10.1111/febs.12253. Epub 2013 Apr 17. PMID 23517348
- [Background] Burd NA, West DW, Staples AW, Atherton PJ, Baker JM, Moore DR, Holwerda AM, Parise G, Rennie MJ, Baker SK, Phillips SM. Low-load high volume resistance exercise stimulates muscle protein synthesis more than high-load low volume resistance exercise in young men. PLoS One. 2010 Aug 9;5(8):e12033. doi: 10.1371/journal.pone.0012033. PMID 20711498
- [Background] Chen L, Nelson DR, Zhao Y, Cui Z, Johnston JA. Relationship between muscle mass and muscle strength, and the impact of comorbidities: a population-based, cross-sectional study of older adults in the United States. BMC Geriatr. 2013 Jul 16;13:74. doi: 10.1186/1471-2318-13-74. PMID 23865675
- [Background] Terzis G, Georgiadis G, Stratakos G, Vogiatzis I, Kavouras S, Manta P, Mascher H, Blomstrand E. Resistance exercise-induced increase in muscle mass correlates with p70S6 kinase phosphorylation in human subjects. Eur J Appl Physiol. 2008 Jan;102(2):145-52. doi: 10.1007/s00421-007-0564-y. Epub 2007 Sep 14. PMID 17874120
- [Background] Tipton KD, Ferrando AA, Phillips SM, Doyle D Jr, Wolfe RR. Postexercise net protein synthesis in human muscle from orally administered amino acids. Am J Physiol. 1999 Apr;276(4):E628-34. doi: 10.1152/ajpendo.1999.276.4.E628. PMID 10198297
- [Background] Srednicka-Tober D, Baranski M, Seal C, Sanderson R, Benbrook C, Steinshamn H, Gromadzka-Ostrowska J, Rembialkowska E, Skwarlo-Sonta K, Eyre M, Cozzi G, Krogh Larsen M, Jordon T, Niggli U, Sakowski T, Calder PC, Burdge GC, Sotiraki S, Stefanakis A, Yolcu H, Stergiadis S, Chatzidimitriou E, Butler G, Stewart G, Leifert C. Composition differences between organic and conventional meat: a systematic literature review and meta-analysis. Br J Nutr. 2016 Mar 28;115(6):994-1011. doi: 10.1017/S0007114515005073. Epub 2016 Feb 16. PMID 26878675
- [Background] Davis H, Magistrali A, Butler G, Stergiadis S. Nutritional Benefits from Fatty Acids in Organic and Grass-Fed Beef. Foods. 2022 Feb 23;11(5):646. doi: 10.3390/foods11050646. PMID 35267281